CLINICAL TRIAL: NCT05868434
Title: Medial Patellofemoral Ligament Reconstruction (MPFLR) With Fascia Lata Allograft, Based on Isometry Assessment Combined With Elmslie-Trillat Tibial Tuberosity Osteotomy.
Brief Title: MPFLR With Fascia Lata Allograft, Based on Isometry Assessment + Elmslie-Trillat TTO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Artromedical Konrad Malinowski Clinic (Other)
Responsible Party: Principal Investigator, Konrad Malinowski MD, Konrad Malinowski MD, Director of Artromedical Konrad Malinowski Clinic and Principal Investigator, Artromedical Konrad Malinowski Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3-pro-ar-2023
Record Dates: First submitted 2023-05-08; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Lateral Patellofemoral Dislocation Closed Traumatic; Lateral Patellar Luxation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Main arm of the study (Experimental): Medial Patellofemoral Ligament Reconstruction (MPFLR) With Fascia Lata Allograft, Based on Isometry Assessment Combined With Elmslie-Trillat Tibial Tuberosity Osteotomy will be performed in these patients.
  Interventions: Procedure: Medial Patellofemoral Ligament Reconstruction (MPFLR) With Fascia Lata Allograft, Based on Isometry Assessment Combined With Elmslie-Trillat Tibial Tuberosity Osteotomy.

INTERVENTIONS:
Procedure: Medial Patellofemoral Ligament Reconstruction (MPFLR) With Fascia Lata Allograft, Based on Isometry Assessment Combined With Elmslie-Trillat Tibial Tuberosity Osteotomy. — Medial Patellofemoral Ligament Reconstruction (MPFLR) With Fascia Lata Allograft, Based on Isometry Assessment Combined With Elmslie-Trillat Tibial Tuberosity Osteotomy. Management of any accompanying patellofemoral lesions will be performed as well.

SUMMARY:
The aim of this study is to assess outcomes of MPFLR With Fascia Lata Allograft, Based on Isometry Assessment Combined With Elmslie-Trillat Tibial Tuberosity Osteotomy.

DETAILED DESCRIPTION:
Medial Patellofemoral Ligament (MPFL) injury occurs in more than 95% of lateral patellar dislocations. Most of these injuries result in subsequent lateral patellar instability. Therefore, MPFL reconstruction (MPFLR) is often necessary. The aim of this study is to assess outcomes of MPFLR With Fascia Lata Allograft, Based on Isometry Assessment Combined With Elmslie-Trillat Tibial Tuberosity Osteotomy.

The primary outcome consists of The International Knee Documentation Committee Questionnaire (IKDC), the Knee injury and Osteoarthritis Outcome Score (KOOS) and retear rate.

ELIGIBILITY:
Inclusion Criteria:

* Lateral patellar dislocation with subsequent instability
* Failure of non-operative treatment

Exclusion Criteria:

* Active inflammation of the knee;
* Previous surgeries on the patellofemoral joint;
* Fractures around the knee

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-02-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Lateral patella stability - apprehension test | At the 12 month of the follow-up.
  Apprehension test at 30 degrees of knee flexion
Lateral patella stability - lateral luxation test | At the 12 month of the follow-up.
  Lateral luxation test at 30 degrees of knee flexion
Lateral patella stability - apprehension test | At the 24 month of the follow-up.
  Apprehension test at 30 degrees of knee flexion
Lateral patella stability - lateral luxation test | At the 24 month of the follow-up.
  Lateral luxation test at 30 degrees of knee flexion

SECONDARY OUTCOMES:
The functional assessment with the The International Knee Documentation Committee Questionnaire (IKDC) | At the 12 month of the follow-up.
  Min of 0 max of 87 points, higher scores mean a better outcome
The functional assessment with the The International Knee Documentation Committee Questionnaire (IKDC) | At the 24 month of the follow-up.
  Min of 0 max of 87 points, higher scores mean a better outcome
The functional assessment with the Knee injury and Osteoarthritis Outcome Score | At the 12 month of the follow-up.
  Min of 0 max of 100 points, higher scores mean a better outcome
The functional assessment with the Knee injury and Osteoarthritis Outcome Score | At the 24 month of the follow-up.
  Min of 0 max of 100 points, higher scores mean a better outcome
ROM | At the 12 month of the follow-up.
  Knee range of motion assessed by the means of goniometer.
ROM | At the 24 month of the follow-up.
  Knee range of motion assessed by the means of goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Konrad Malinowski, MD PhD, Principal Investigator — Artromedical Orthopaedic Clinic, Bełchatów, Poland
Locations (1):
- Artromedical Orthopaedic Clinic, Bełchatów, Łódź Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ryan PC, Ross BJ, Stamm MA, Sherman WF, Heard WMR, Mulcahey MK. Concomitant Tibial Tubercle Osteotomy Reduces the Risk of Revision Surgery After Medial Patellofemoral Ligament Reconstruction for the Treatment of Patellar Instability. Arthroscopy. 2023 Sep;39(9):2037-2045.e1. doi: 10.1016/j.arthro.2023.02.006. Epub 2023 Feb 18. PMID 36804459
- [Background] Agarwalla A, Gowd AK, Liu JN, Puzzitiello RN, Yanke AB, Verma NN, Forsythe B. Concomitant Medial Patellofemoral Ligament Reconstruction and Tibial Tubercle Osteotomy Do Not Increase the Incidence of 30-Day Complications: An Analysis of the NSQIP Database. Orthop J Sports Med. 2019 Apr 12;7(4):2325967119837639. doi: 10.1177/2325967119837639. eCollection 2019 Apr. PMID 31019984
- [Background] Franciozi CE, Ambra LF, Albertoni LJB, Debieux P, Granata GSM Jr, Kubota MS, Carneiro M, Abdalla RJ, Luzo MVM, Cohen M. Anteromedial Tibial Tubercle Osteotomy Improves Results of Medial Patellofemoral Ligament Reconstruction for Recurrent Patellar Instability in Patients With Tibial Tuberosity-Trochlear Groove Distance of 17 to 20 mm. Arthroscopy. 2019 Feb;35(2):566-574. doi: 10.1016/j.arthro.2018.10.109. Epub 2019 Jan 4. PMID 30612771
- [Background] Aliberti GM, Kraeutler MJ, Miskimin C, Scillia AJ, Belk JW, Mulcahey MK. Autograft Versus Allograft for Medial Patellofemoral Ligament Reconstruction: A Systematic Review. Orthop J Sports Med. 2021 Oct 19;9(10):23259671211046639. doi: 10.1177/23259671211046639. eCollection 2021 Oct. PMID 34692883
- [Background] Allen MM, Krych AJ, Johnson NR, Mohan R, Stuart MJ, Dahm DL. Combined Tibial Tubercle Osteotomy and Medial Patellofemoral Ligament Reconstruction for Recurrent Lateral Patellar Instability in Patients With Multiple Anatomic Risk Factors. Arthroscopy. 2018 Aug;34(8):2420-2426.e3. doi: 10.1016/j.arthro.2018.02.049. Epub 2018 May 19. PMID 29789255
- [Background] Lobner S, Krauss C, Reichwein F, Patzer T, Nebelung W, Venjakob AJ. Surgical treatment of patellar instability: clinical and radiological outcome after medial patellofemoral ligament reconstruction and tibial tuberosity medialisation. Arch Orthop Trauma Surg. 2017 Aug;137(8):1087-1095. doi: 10.1007/s00402-017-2705-z. Epub 2017 May 16. PMID 28508959